CLINICAL TRIAL: NCT05445531
Title: Low-field Magnetic Resonance Imaging to Assess Changes in Pulmonary Function Parameters in Confirmed Pediatric SARS-CoV-2 Infection
Brief Title: Low-field Magnetic Resonance Imaging in Pediatric Post Covid-19
Acronym: FASCINATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-77-Bm
Record Dates: First submitted 2022-07-05; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: COVID-19; COVID-19 Respiratory Infection; Long COVID
Keywords: COVID-19; Long COVID; post COVID
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Microscopic Angioscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Proof of SARS-CoV-2 infection and at least 2/3 times complete vaccination before infection (at least 14 days) (complete vaccination status according to STIKO, German vaccination committee)
  Interventions: Diagnostic Test: Low-field magnetic resonance imaging; Diagnostic Test: Nailfold capillaroscopy; Diagnostic Test: Spiroergometry; Diagnostic Test: Realtime deformability cytometry
- Recovered (Active Comparator): Positive SARS-CoV-2 infection confirmed by PCR; Long Covid criteria according to AWMF S1 guideline not fulfilled.
  Interventions: Diagnostic Test: Low-field magnetic resonance imaging; Diagnostic Test: Nailfold capillaroscopy; Diagnostic Test: Spiroergometry; Diagnostic Test: Realtime deformability cytometry
- Long Covid (Experimental): Positive SARS-CoV-2 infection confirmed by PCR; Long Covid criteria according to AWMF S1 guideline fulfilled.
  Interventions: Diagnostic Test: Low-field magnetic resonance imaging; Diagnostic Test: Nailfold capillaroscopy; Diagnostic Test: Spiroergometry; Diagnostic Test: Realtime deformability cytometry

INTERVENTIONS:
Diagnostic Test: Low-field magnetic resonance imaging — Functional and morphologic imaging of the lungs
  Other Names: LF-MRI
Diagnostic Test: Nailfold capillaroscopy — Imaging of nailfold microvasculature
Diagnostic Test: Spiroergometry — Cardiopulmonary exercise testing
Diagnostic Test: Realtime deformability cytometry — High-throughput measurement of cell deformability and physical properties
  Other Names: RT-DC

SUMMARY:
SARS-CoV-2 (Severe acute respiratory syndrome coronavirus type 2) is a new coronavirus and identified causative agent of COVID-19 disease. These viruses predominantly cause mild colds, but can sometimes cause severe pneumonia and pulmonary skeletal changes. By low-field gastric magnetic resonance imaging (NF-MRI), only a small number of structural, scarring changes were seen in a preliminary study of pediatric and adolescent patients with past SARS-CoV-2 infection. In contrast, however, extensive changes in ventilation and blood flow function of the lungs were seen.

The long-term consequences and spontaneous progression of these changes on imaging are completely unclear. The aim of this study is to assess the course of these functional lung changes in pediatric and adolescent patients and to validate them with other standard clinical procedures.

DETAILED DESCRIPTION:
SARS-CoV-2 (Severe acute respiratory syndrome coronavirus type 2) is a new coronavirus and identified causative agent of COVID-19 disease. They predominantly cause mild colds but can sometimes cause severe pneumonia and pulmonary skeletal disease. While the molecular basis for the changes in lung tissue or multi-organ involvement have been described, the age-specific long-term consequences, especially in children and adolescents, remain largely unexplained and misunderstood today.

Early publications from the primarily affected Chinese provinces described rather mild, partly asymptomatic courses in children. This is consistent with the observation that the risk of severe COVID-19 disease increases steeply from the age of 70 years, and is also determined by the severity of obesity as well as other risk factors. Developmental expression of tissue factors may be one reason for the relative protection of younger patients from severe courses of the disease.

However, it is now becoming increasingly clear that some individuals with milder initial symptoms of COVID-19 may suffer from variable and persistent symptoms for many months after initial infection - this includes children. A modern low-field MRI is located in Erlangen, Germany. This technique has already been used to demonstrate persistent damage to lung tissue in adult patients after COVID-19. The device with a field strength of 0.55 Tesla (T) currently has the world's largest aperture (and is thus particularly suitable for patients with claustrophobia, among other things), a very quiet operating noise, and lower energy absorption in the tissue due to the weaker magnetic field than MRI scanners with 1.5T or 3T. This allows MRI imaging in a very broad pediatric population without the need for sedation.

To date, no structural changes were revealed by means of this MRI technique - however, large defects in the area of ventilation and blood flow function of the lung are apparent in specific functional sequences. The aim of this study is to assess the course of these functional lung changes in pediatric and adolescent patients and to validate them with other standard clinical procedures.

ELIGIBILITY:
Control arm:

Inclusion Criteria:

* Proof of SARS-CoV-2 infection and at least 2/3 times complete vaccination before infection (at least 14 days) (complete vaccination status according to German recommendations)
* Long Covid criteria not met according to AWMF S1 guideline

Exclusion Criteria:

* Acute SARS-CoV-2 infection and need for isolation
* Necessary quarantine
* Pregnancy, lactation
* Indication of acute infection
* Known pleural or pericardial effusion
* Critical condition (need for respiratory support, ventilation, oxygen administration, shock, symptomatic heart failure)
* Marked thoracic deformities
* Previous lung surgery
* Injuries that do not allow for physical stress testing
* Refusal of MRI imaging
* General contraindications to MRI examinations (e.g., electrical implants such as pacemakers or perfusion pumps, etc.)
* History, clinical, or other suspicion of pulmonary disease
* Current respiratory infection/symptomatology
* Pain leading to respiratory limitation
* Inhaled therapy (e.g., steroids or beta-mimetics)
* Immunosuppression
* Any condition that may lead to respiratory limitation (e.g., pain disorder)
* Obesity (>97% of age percentile)

Recovered arm:

Inclusion Criteria:

* Positive SARS-CoV-2 infection confirmed by PCR
* Long Covid criteria not met according to AWMF S1 guideline

Exclusion Criteria:

* Acute SARS-CoV-2 infection and need for isolation
* Necessary quarantine
* Pregnancy, lactation
* Indication of acute infection
* Known pleural or pericardial effusion
* Critical condition (need for respiratory support, ventilation, oxygen administration, shock, symptomatic heart failure)
* Marked thoracic deformities
* Previous lung surgery
* Injuries that do not allow for physical stress testing
* Refusal of MRI imaging
* General contraindications to MRI examinations (e.g., electrical implants such as pacemakers or perfusion pumps, etc.)

Long Covid arm:

Inclusion Criteria:

* Positive SARS-CoV-2 infection confirmed by PCR
* Long Covid criteria according to AWMF S1 guideline fulfilled

Exclusion Criteria:

* Acute SARS-CoV-2 infection and need for isolation
* Necessary quarantine
* Pregnancy, lactation
* Indication of acute infection
* Known pleural or pericardial effusion
* Critical condition (need for respiratory support, ventilation, oxygen administration, shock, symptomatic heart failure)
* Marked thoracic deformities
* Previous lung surgery
* Injuries that do not allow for physical stress testing
* Refusal of MRI imaging
* General contraindications to MRI examinations (e.g., electrical implants such as pacemakers or perfusion pumps, etc.)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Estimated)
Dates: Start 2022-07-08 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Functional lung assessment (LF-MRI) | Baseline compared to 6 months
  Change in functional lung parameters

SECONDARY OUTCOMES:
Morphologic lung assessment (LF-MRI) | Baseline compared to 6 months
  Morphologic changes in lung parenchyma
Cardiological functional diagnostics (VO2) | Baseline compared to 6 months
  Oxygen uptake (VO2)
Cardiological functional diagnostics (VO2max) | Baseline compared to 6 months
  Peak oxygen uptake (VO2max)
Cardiological functional diagnostics (VT2) | Baseline compared to 6 months
  Ventilatory anaerobic threshold (VT2)
Cardiological functional diagnostics (VCO2) | Baseline compared to 6 months
  Carbon dioxide output (VCO2)
Cardiological functional diagnostics (HR) | Baseline compared to 6 months
  Heart rate (HR)
Cardiological functional diagnostics (HRR) | Baseline compared to 6 months
  Heart Rate Reserve (HRR)
Cardiological functional diagnostics (Breath rate at VAT) | Baseline compared to 6 months
  Breath rate at VAT
Cardiological functional diagnostics (BRR) | Baseline compared to 6 months
  Breath rate reserve (BRR)
Cardiological functional diagnostics (VE) | Baseline compared to 6 months
  Minute ventilation (VE)
Cardiological functional diagnostics (O2Pulse) | Baseline compared to 6 months
  O2Pulse
Cardiological functional diagnostics (HRV) | Baseline compared to 6 months
  Heart rate variability (HRV)
Cardiological functional diagnostics (Borg Scale) | Baseline compared to 6 months
  Exercise capacity nach Borg Scale
Cardiological functional diagnostics (BGA) | Baseline compared to 6 months
  Capillary blood gas and lactate (BGA)
Nailfold capillaroscopy (capillaries) | Baseline compared to 6 months
  Number of capillaries in first row
Nailfold capillaroscopy (first row) | Baseline compared to 6 months
  Number of capillaries in first row
Nailfold capillaroscopy (morphology) | Baseline compared to 6 months
  Morphology of capillaries
Blood sample (antibodies) | Baseline compared to 6 months
  SARS-CoV2-antibodies
Blood sample (auto antibodies) | Baseline compared to 6 months
  Autoantibodies against G-protein receptors
Blood sample (RT-DC) | Baseline compared to 6 months
  Realtime deformability cytometry
Blood sample (Blood count) | Baseline compared to 6 months
  Blood count
Blood sample (IL-6) | Baseline compared to 6 months
  Interleukin-6 (IL-6)
Blood sample (CrP) | Baseline compared to 6 months
  C-reactive proteine (CrP)
Blood sample (Calpro) | Baseline compared to 6 months
  Calprotectin (Calpro)
Blood sample (Coagulation) | Baseline compared to 6 months
  Coagulation factors (Coagulation)

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinand Knieling, MD, Principal Investigator — University Hospital Erlangen
Locations (1):
- University Hospital Erlangen, Erlangen, Bavaria, Germany

REFERENCES:
- [Background] Sajuthi SP, DeFord P, Li Y, Jackson ND, Montgomery MT, Everman JL, Rios CL, Pruesse E, Nolin JD, Plender EG, Wechsler ME, Mak ACY, Eng C, Salazar S, Medina V, Wohlford EM, Huntsman S, Nickerson DA, Germer S, Zody MC, Abecasis G, Kang HM, Rice KM, Kumar R, Oh S, Rodriguez-Santana J, Burchard EG, Seibold MA. Type 2 and interferon inflammation regulate SARS-CoV-2 entry factor expression in the airway epithelium. Nat Commun. 2020 Oct 12;11(1):5139. doi: 10.1038/s41467-020-18781-2. PMID 33046696
- [Background] Ziegler CGK, Allon SJ, Nyquist SK, Mbano IM, Miao VN, Tzouanas CN, Cao Y, Yousif AS, Bals J, Hauser BM, Feldman J, Muus C, Wadsworth MH 2nd, Kazer SW, Hughes TK, Doran B, Gatter GJ, Vukovic M, Taliaferro F, Mead BE, Guo Z, Wang JP, Gras D, Plaisant M, Ansari M, Angelidis I, Adler H, Sucre JMS, Taylor CJ, Lin B, Waghray A, Mitsialis V, Dwyer DF, Buchheit KM, Boyce JA, Barrett NA, Laidlaw TM, Carroll SL, Colonna L, Tkachev V, Peterson CW, Yu A, Zheng HB, Gideon HP, Winchell CG, Lin PL, Bingle CD, Snapper SB, Kropski JA, Theis FJ, Schiller HB, Zaragosi LE, Barbry P, Leslie A, Kiem HP, Flynn JL, Fortune SM, Berger B, Finberg RW, Kean LS, Garber M, Schmidt AG, Lingwood D, Shalek AK, Ordovas-Montanes J; HCA Lung Biological Network. Electronic address: lung-network@humancellatlas.org; HCA Lung Biological Network. SARS-CoV-2 Receptor ACE2 Is an Interferon-Stimulated Gene in Human Airway Epithelial Cells and Is Detected in Specific Cell Subsets across Tissues. Cell. 2020 May 28;181(5):1016-1035.e19. doi: 10.1016/j.cell.2020.04.035. Epub 2020 Apr 27. PMID 32413319
- [Background] Huang J, Hume AJ, Abo KM, Werder RB, Villacorta-Martin C, Alysandratos KD, Beermann ML, Simone-Roach C, Lindstrom-Vautrin J, Olejnik J, Suder EL, Bullitt E, Hinds A, Sharma A, Bosmann M, Wang R, Hawkins F, Burks EJ, Saeed M, Wilson AA, Muhlberger E, Kotton DN. SARS-CoV-2 Infection of Pluripotent Stem Cell-Derived Human Lung Alveolar Type 2 Cells Elicits a Rapid Epithelial-Intrinsic Inflammatory Response. Cell Stem Cell. 2020 Dec 3;27(6):962-973.e7. doi: 10.1016/j.stem.2020.09.013. Epub 2020 Sep 18. PMID 32979316
- [Background] Karki R, Sharma BR, Tuladhar S, Williams EP, Zalduondo L, Samir P, Zheng M, Sundaram B, Banoth B, Malireddi RKS, Schreiner P, Neale G, Vogel P, Webby R, Jonsson CB, Kanneganti TD. Synergism of TNF-alpha and IFN-gamma Triggers Inflammatory Cell Death, Tissue Damage, and Mortality in SARS-CoV-2 Infection and Cytokine Shock Syndromes. Cell. 2021 Jan 7;184(1):149-168.e17. doi: 10.1016/j.cell.2020.11.025. Epub 2020 Nov 19. PMID 33278357
- [Background] Lu X, Zhang L, Du H, Zhang J, Li YY, Qu J, Zhang W, Wang Y, Bao S, Li Y, Wu C, Liu H, Liu D, Shao J, Peng X, Yang Y, Liu Z, Xiang Y, Zhang F, Silva RM, Pinkerton KE, Shen K, Xiao H, Xu S, Wong GWK; Chinese Pediatric Novel Coronavirus Study Team. SARS-CoV-2 Infection in Children. N Engl J Med. 2020 Apr 23;382(17):1663-1665. doi: 10.1056/NEJMc2005073. Epub 2020 Mar 18. No abstract available. PMID 32187458
- [Background] Brodin P. Immune determinants of COVID-19 disease presentation and severity. Nat Med. 2021 Jan;27(1):28-33. doi: 10.1038/s41591-020-01202-8. Epub 2021 Jan 13. PMID 33442016
- [Background] Schuler BA, Habermann AC, Plosa EJ, Taylor CJ, Jetter C, Negretti NM, Kapp ME, Benjamin JT, Gulleman P, Nichols DS, Braunstein LZ, Hackett A, Koval M, Guttentag SH, Blackwell TS, Webber SA, Banovich NE; Vanderbilt COVID-19 Consortium Cohort; Human Cell Atlas Biological Network; Kropski JA, Sucre JM. Age-determined expression of priming protease TMPRSS2 and localization of SARS-CoV-2 in lung epithelium. J Clin Invest. 2021 Jan 4;131(1):e140766. doi: 10.1172/JCI140766. PMID 33180746
- [Background] Heiss R, Grodzki DM, Horger W, Uder M, Nagel AM, Bickelhaupt S. High-performance low field MRI enables visualization of persistent pulmonary damage after COVID-19. Magn Reson Imaging. 2021 Feb;76:49-51. doi: 10.1016/j.mri.2020.11.004. Epub 2020 Nov 18. PMID 33220447
- [Background] Shelmerdine SC, Lovrenski J, Caro-Dominguez P, Toso S; Collaborators of the European Society of Paediatric Radiology Cardiothoracic Imaging Taskforce. Coronavirus disease 2019 (COVID-19) in children: a systematic review of imaging findings. Pediatr Radiol. 2020 Aug;50(9):1217-1230. doi: 10.1007/s00247-020-04726-w. Epub 2020 Jun 18. PMID 32556807
- [Background] Duan YN, Zhu YQ, Tang LL, Qin J. CT features of novel coronavirus pneumonia (COVID-19) in children. Eur Radiol. 2020 Aug;30(8):4427-4433. doi: 10.1007/s00330-020-06860-3. Epub 2020 Apr 14. PMID 32291501
- [Background] Steinberger S, Lin B, Bernheim A, Chung M, Gao Y, Xie Z, Zhao T, Xia J, Mei X, Little BP. CT Features of Coronavirus Disease (COVID-19) in 30 Pediatric Patients. AJR Am J Roentgenol. 2020 Dec;215(6):1303-1311. doi: 10.2214/AJR.20.23145. Epub 2020 May 22. PMID 32442030
- [Derived] Weigelt A, Akhundova G, Raming R, Tratzky JP, Regensburger AP, Kraus C, Waellisch W, Trollmann R, Woelfle J, Dittrich S, Heiss R, Knieling F, Schoeffl I. Light at the end of the tunnel? Follow-up of cardiopulmonary function in children with post-COVID-19. Eur J Pediatr. 2025 Jun 10;184(7):413. doi: 10.1007/s00431-025-06245-y. PMID 40495009